CLINICAL TRIAL: NCT06105229
Title: Clinical Value of Plasma Humanin in Acute Kidney Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Li zhilian, Deputy Chief Physician, Guangdong Provincial People's Hospital
Other Study IDs: NO.GDREC2020278H
Record Dates: First submitted 2023-10-07; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute kidney injury: Patients with AKI who meet KDIGO criteria
- Healthy controls: Healthy people without other underlying medical conditions

SUMMARY:
The goal of this observational study is to assess the clinical value of humanin in acute kidney injury. The main questions it aims to answer are:whether Humanin can be a novel marker for predicting AKI Researchers will compare humanin concentration in healthy people to see if humanin can be a novel marker for predicting AKI

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI) is a clinically critical condition manifested by a sharp decline in kidney function, with approximately 13.3 million people diagnosed with AKI each year in hospital worldwide and associated with 1.7 million deaths. According to global multi-center research data, the total incidence of AKI in hospital is as high as 21%, and the incidence of acute kidney injury in hospitalized patients in China is 0.99%~11.6%. AKI increases the risk of long-term chronic kidney disease (CKD) and end-stage renal disease (ESRD), and has a very high long-term mortality rate. The diagnosis of AKI is mainly based on blood creatinine or urine output, and the current KDIGO criteria are used, but blood creatinine is a very insensitive indicator, so in the past 20 years, scholars have been exploring biological markers that are more sensitive than blood creatinine and urine output. Humanin is a mitochondrial polypeptide containing 24 amino acids. It was first identified in Alzheimer's disease patients in 2001. Studies have shown that Humanin has a strong mitochondrial protective effect in neurodegenerative diseases, cardiovascular diseases, diabetes, male infertility, cancer and other diseases, and its mechanism may be related to anti-apoptosis, anti-inflammation, regulation of autophagy and maintenance of mitochondrial homeostasis, because Humanin can function through autocrine, paracrine or endocrine forms, so it can be detected in the blood. Studies have shown that Humanin expression in serum or plasma of patients with diabetes and coronary heart disease is declined. In our previous study, the investigators found that Humanin was elevated in plasma in a mouse model of AKI with sepsis.

The goal of this observational study is to assess the clinical value of humanin in acute kidney injury. The main questions it aims to answer are:whether Humanin can be a novel marker for predicting AKI

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age, male or female；
* Patients with AKI: Patients with acute kidney injury who meet the definition of KDIGO guidelines；
* Control group: from healthy physical examination population, physical examination blood routine, urine routine, liver function, kidney function, glycated hemoglobin and other indicators are normal；
* The patient's baseline medical record data is complete, including liver and kidney function, urine protein level, blood creatinine value, etc；
* Consent to enrollment and sign informed consent；

Exclusion Criteria:

* Age< 18 years；
* Baseline data were missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AKI patients from Guangdong Provincial People's Hospital from 2023 to May 2024
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Humanin concentration | one week
  Highest measured value used
Serum creatinine concentration | one week
  Meets KDIGO's definition of AKI

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangdong, Guangzhou, China

DOCUMENTS (1):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT06105229/Prot_000.pdf